CLINICAL TRIAL: NCT02509858
Title: The Effect of Administration of Small Doses of Thyroxine on Glucose and Lipid Metabolism, at All Stages of Type 2 Diabetes Mellitus.
Brief Title: The Effect of Administration of Small Doses of Thyroxine on Glucose and Lipid Metabolism, in Type 2 Diabetes Mellitus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Assistant Professor of of Internal Medicine and Clinical Diabetology , University of Athens, Greece, Attikon Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ΒΠΠΚ 50/11-02-09
Record Dates: First submitted 2015-07-26; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus, thyroxine
MeSH Terms: conditions — Diabetes Mellitus | interventions — Thyroxine; CD36 Antigens; Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- thyroxine in eythyroid diabetics (Active Comparator): 50 μg of thyroxine once daily, for 2 months.
  Interventions: Drug: thyroxine; Other: A meal (730kcal, 50%carbohydrate, of which 38% was starch, 40% fat, and 10% protein)
- thyroxine in euthyroid healthy humans (Active Comparator): 50 μg of thyroxine once daily, for 2 months.
  Interventions: Drug: thyroxine; Other: A meal (730kcal, 50%carbohydrate, of which 38% was starch, 40% fat, and 10% protein)
- placebo in euthyroid diabetics (Placebo Comparator): 50 μg of placebo once daily, for 2 months.
  Interventions: Drug: Placebo; Other: A meal (730kcal, 50%carbohydrate, of which 38% was starch, 40% fat, and 10% protein)

INTERVENTIONS:
Drug: thyroxine — treatment with 50μg of thyroxine once daily for two months.
  Other Names: T4
  Arms: thyroxine in euthyroid healthy humans; thyroxine in eythyroid diabetics
Drug: Placebo — treatment with 50μg of placebo, once daily, for two months.
  Arms: placebo in euthyroid diabetics
Other: A meal (730kcal, 50%carbohydrate, of which 38% was starch, 40% fat, and 10% protein)

SUMMARY:
We investigated the effect of the administration of small doses of thyroxine to healthy humans and patients with type 2 diabetes on postprandial forearm muscle glucose uptake, insulin sensitivity indices, lipid metabolism, in vitro glucose uptake and GLUT4 recruitment in the plasma membrane of monocytes.

DETAILED DESCRIPTION:
The present open-labeled, randomized and placebo-controlled study was undertaken in euthyroid type 2 diabetic patients and healthy humans, to examine the effect of administration of small doses of thyroxine within the euthyroid range, on muscle glucose disposal, postprandial insulin sensitivity, lipid metabolism, in vitro glucose uptake and GLUT4 recruitment in the plasma membrane of monocytes.This was investigated with the arteriovenous-difference technique after the consumption of a mixed meal and the in vitro study of a glucose analogue(6-NBDG) uptake by the peripheral monocytes.

Subjects and Methods: Eleven euthyroid, treatment naive, type-2 diabetic patients with a micronodular texture of the thyroid gland and eleven healthy euthyroid subjects, were studied before and after administration of 50 μg of thyroxine once daily for 2 months. In parallel, a placebo group was also studied. Eleven euthyroid treatment-naïve subjects with type 2 diabetes and a micronodular texture of the thyroid gland, matched for age, sex, BMI, and basal thyroid function, were studied before and after administration of a placebo, once daily for 2 months.

Experimental protocol: All subjects were admitted to the hospital at 0700 h after an overnight fast and had the radial artery (A) and a forearm deep vein (V) catheterized. A meal (730kcal, 50%carbohydrate, of which 38% was starch, 40% fat, and 10% protein) was given at least 1 h after catheter insertion and was consumed within 20 min. Blood samples were drawn from both sites before the meal (at -30 and 0 min) and at 30- to 60-min intervals for 300 min thereafter for measurements of thyroid hormones,glucose, total cholesterol, LDL Cholesterol, HDL Cholesterol, triglycerides, Apolipoprotein A1, Apolipoprotein BII and Lp(a).Forearm blood flow was measured with strain-gauge plethysmography. After the first meal tolerance test, treatment with 50μg of thyroxine or placebo, once daily, was initiated for a 2-month period. Then a second identical test was repeated. Special care was taken in order to avoid the induction of subclinical hyperthyroidism, that is suppression of TSH below 0.27 μU/ml, as it has recently been shown that the latter is also an insulin-resistant condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or treatment naive type 2 diabetes euthyroid subjects, with a micronodular texture of the thyroid gland.
* Recreationally active
* With stable body weight and diet during the last two months.

Exclusion Criteria:

* Any systemic disease(besides glucose abnormalities)
* Any medication therapy
* Diabetic complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-02; Primary Completion 2014-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
area under the glucose uptake versus time curve-AUC | Time Frame: 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  Muscle glucose uptake following meal ingestion

SECONDARY OUTCOMES:
Plasma glucose levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma insulin levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma triglyceride levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma total cholesterol levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma LDL-cholesterol levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma HDL-cholesterol levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma Apo-A levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma Apo-B levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma Lp(α) levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma NEFA levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma glycerol levels following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Muscle blood flow following meal ingestion | 0, 30, 60, 90, 120, 180, 240, 300 min postmeal
  area under the plasma concentration versus time curve-AUC
Plasma thyroid hormones | baseline
  measure of plasma concentration
glucose uptake by peripheral monocytes by the usage of the fluorescent analogue 6-NBDG | baseline to 600 sec
  area under the curve of 6-NBDG uptake by monocytes under insulin stimulation
% GLUT4 increment from baseline (0mU/l) to maximal concentration (200mU/l) of insulin. | baseline
Number of participants with adverse events | 300 min postmeal

CONTACTS AND LOCATIONS:
Overall Officials: GEORGE DIMITRIADIS, MD, Phd, Study Director — 2nd Department of Internal Medicine, Research Institute and Diabetes Center, Athens University Medical School, Attikon Hospital